CLINICAL TRIAL: NCT01884116
Title: Comparison of NSAID Patch Given in Monotherapy and NSAID Patch in Combination With Transcutaneous Electric Nerve Stimulation, Heating Pad, or Topical Capsaicin in the Treatment of Patients With Myofascial Pain Syndrome of the Upper Trapezius: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1-2010-0060
Record Dates: First submitted 2013-06-14; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Myofascial Pain Syndrome of the Upper Trapezius
Keywords: Capsaicin; myofascial pain syndrome; non-steroidal anti-inflammatory agents; transcutaneous electric nerve stimulation
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Transcutaneous Electric Nerve Stimulation; Capsaicin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NSAID patch group (Active Comparator): administer the NSAID patch
  Interventions: Drug: NSAID patch
- NSAID patch + transcutaneous electric nerve stimulation group (Experimental)
  Interventions: Drug: NSAID patch + transcutaneous electric nerve stimulation
- NSAID patch + heating pad group (Experimental)
  Interventions: Drug: NSAID patch + heating pad
- NSAID patch + topical capsaicin group (Experimental)
  Interventions: Drug: NSAID patch + topical capsaicin

INTERVENTIONS:
Drug: NSAID patch
  Arms: NSAID patch group
Drug: NSAID patch + transcutaneous electric nerve stimulation — The patients of the experimental groups will be divided in to three groups according to what they are administered: NSAID patch plus transcutaneous electric nerve stimulation, NSAID patch plus heating pad, and NSAID patch plus topical capsaicin. All the groups will be observed for two weeks.
  Arms: NSAID patch + transcutaneous electric nerve stimulation group
Drug: NSAID patch + heating pad — The patients of the experimental groups will be divided in to three groups according to what they are administered: NSAID patch plus transcutaneous electric nerve stimulation, NSAID patch plus heating pad, and NSAID patch plus topical capsaicin. All the groups will be observed for two weeks.
  Arms: NSAID patch + heating pad group
Drug: NSAID patch + topical capsaicin — The patients of the experimental groups will be divided in to three groups according to what they are administered: NSAID patch plus transcutaneous electric nerve stimulation, NSAID patch plus heating pad, and NSAID patch plus topical capsaicin. All the groups will be observed for two weeks.
  Arms: NSAID patch + topical capsaicin group

SUMMARY:
Myofascial pain syndrome (MPS) is a common clinical problem of musculoskeletal pain and various treatment modalities have been introduced. If self-applicable physical modalities and medications that are used for treatment of MPS patients are combined, they may open up new possibilities for effective and practical self-care. The aim of this study is to compared the therapeutic effect of non-steroidal anti-inflammatory drug (NSAID) patch given in monotherapy and NSAID patch in combination with transcutaneous electric nerve stimulation, heating pad, or topical capsaicin in the treatment of patients with MPS of the upper trapezius.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 20 years of age with diagnosis of myofascial pain syndrome of the upper trapezius.
2. Visual analogue scale (VAS, 0 = no pain, 10 = worst pain) greater than

Exclusion Criteria:

1. Pregnant or breast feeding women, patients who have taken opioids within seven days, patients with severe disease (heart disease, liver disease, etc) that might affect the results of the study, patients who have participated in another clinical study within 30 days.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The differences of the VAS pain scores | 2weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Al-Shaikh B, George William M, Van Zundert AA. Using atmospheric pressure to inflate the cuff of the Portex Laryngeal Mask. Anaesthesia. 2005 Mar;60(3):296-7. doi: 10.1111/j.1365-2044.2005.04135.x. No abstract available. PMID 15710025